CLINICAL TRIAL: NCT06920498
Title: A Multipart Phase 1 Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study With Single and Multiple Dose Escalation to Evaluate the Safety, Tolerability, and Pharmacokinetics of PF-07941944 in Healthy Adult Participants
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07941944 Are Tolerated in the Body of Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5961001; 2024-515421-28-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-12-05; First posted 2025-04-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Respiratory syncytial virus (RSV)
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 (Experimental): Single ascending dose of PF-07941944 or placebo in healthy adult participants
  Interventions: Drug: PF-07941944; Drug: Placebo
- Part 2 (Experimental): Multiple doses of PF-07941944 or placebo in healthy adult participants
  Interventions: Drug: PF-07941944; Drug: Placebo
- Part 3 (Optional) (Experimental): Period 1, single dose of Midazolam. Period 2, multiple doses of PF-07941944 + Midazolam
  Interventions: Drug: PF-07941944; Drug: Midazolam

INTERVENTIONS:
Drug: PF-07941944 — Oral formulation
Drug: Placebo — Oral formulation
  Arms: Part 1; Part 2
Drug: Midazolam — Oral formulation
  Arms: Part 3 (Optional)

SUMMARY:
The purpose of this clinical trial is to learn about the safety and tolerability of the study medicine (called PF-07941944) in healthy participants.

This study is seeking participants who:

* Are male or female between the ages of 18 and 60
* Are generally healthy

The investigators will compare the experiences of people receiving the study medicine to those of the people who do not. This will help the investigators determine if the study medicine is safe and well tolerated.

Participants enrolled in Part 1 will take part in this study for approximately 4 months. Participants enrolled in Part 2 or Part 3 will take part in this study for approximately 2.5 months. Study visits will take place at the study clinic. The study team will also call participants once at the end of the study over the phone.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Body mass index (BMI) of 17.5 to 30.5 kg/m2
* For inclusion of Japanese participants: participants who have 4 Japanese biologic grandparents who were born in Japan.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions that may increase the risk of study participation
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 28 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Part 3 only: History of acute narrow-angle glaucoma, untreated open-angle glaucoma, sleep apnea, respiratory insufficiency, myasthenia gravis, or adverse reaction to midazolam or other benzodiazepines. History of hypersensitivity reaction to midazolam, or any of the formulation components.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
Maximum Observed Plasma Concentration (Cmax) | Baseline through end of study, approximately 16 weeks
  Part 3
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | Baseline through end of study, approximately 16 weeks
  Part 3 - if data permit
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Baseline through end of study, approximately 16 weeks
  Part 3 - If AUCinf not collected

SECONDARY OUTCOMES:
Cmax | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2
AUClast | Baseline through end of study, approximately 16 weeks
  Part 1 - if data permit
AUCinf | Baseline through end of study, approximately 16 weeks
  Part 1 - if data permit
Plasma Decay Half-Life (t1/2) | Baseline through end of study, approximately 16 weeks
  Part 1 and Part 2 - if data permit
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | Baseline through end of study, approximately 16 weeks
  Part 2
Number of Participants With Treatment Emergent Treatment-Related AEs | Baseline through end of study, approximately 16 weeks
  Part 3 - Optional
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline through end of study, approximately 16 weeks
  Part 3 - Optional
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline through end of study, approximately 16 weeks
  Part 3 - Optional
Number of Participants With Change From Baseline in ECG Findings | Baseline through end of study, approximately 16 weeks
  Part 3 - Optional

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5961001